CLINICAL TRIAL: NCT06906120
Title: The Effect of Operating Room Introduction With Virtual Reality Glasses on Anxiety, Surgical Fear, and Satisfaction Levels in Patients Undergoing Orthopedic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Acibadem Altunizade Hospital, Istanbul (Unknown); Acibadem Atasehir Hospital (Other)
Responsible Party: Principal Investigator, Rana Güngör Sevinç, Principal Investigator Rana Güngör Sevinç, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTO2025-VR01
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Artroscopic Surgery; Orthopedic Surgery
Keywords: virtual reality illustration; Orthopedic surgery; Virtual reality; Surgical anxiety; Surgical fear; Preoperative education; Patient satisfaction; Pain management; Physiological parameters; Surgical preparation; VR intervention; Pain assessment; Electrodermal activity; Patient education tools; Preoperative anxiety reduction
MeSH Terms: conditions — Patient Satisfaction; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality-Based Education Group (Experimental)
  Interventions: Behavioral: Virtual Reality-Based Operating Room Education
- Standard Education Group (No Intervention)

INTERVENTIONS:
Behavioral: Virtual Reality-Based Operating Room Education — For the Intervention Group:
  Written informed consent will be obtained one day before surgery when patients visit the anesthesia clinic.
  Subsequently, the Patient Introduction Form, State-Trait Anxiety Inventory (STAI-I, STAI-II), and Surgical Fear Scale will be completed, and electrodermal activity data and physiological parameters will be recorded for 5 minutes.
  Participants will watch a 3D training video created by the researcher using Meta Quest 3 virtual reality headsets. This video will provide an introduction to the operating room environment and related procedures.
  After the video, physiological parameters will be recorded again, and STAI-I and the Surgical Fear Scale will be completed.
  On the day of the surgery, after the patients are admitted and necessary preparations are made, STAI-I and the Surgical Fear Scale will be completed again, and physiological parameters will be recorded.
  Electrodermal activity data will be recorded 15-20 minutes before anesthesia is administ
  Other Names: VR-Based Operating Room Orientation; Virtual Reality Surgical Environment Training
  Arms: Virtual Reality-Based Education Group

SUMMARY:
This study aims to evaluate the effects of an operating room tour conducted using virtual reality (VR) goggles on anxiety, surgical fear, post-operative pain, satisfaction levels, and physiological parameters in patients undergoing orthopedic surgery.

The intervention will involve a 360 degree educational video introducing the operating room environment, surgical team roles, and expected patient experience during the perioperative period. This video will be presented using Meta Quest 3 VR goggles. Participants in the intervention group will watch this video before surgery, while the control group will receive standard preoperative education.

The primary outcomes include changes in preoperative anxiety (STAI-I), surgical fear (Surgical Fear Scale), and physiological parameters (e.g., heart rate, blood pressure, and electrodermal activity). Secondary outcomes include post-operative pain and patient satisfaction. Data will be collected at multiple time points, including before and after the intervention, on the day of surgery, and during the postoperative period.

The study is designed as a randomized controlled trial with a sample size of 60 participants, equally distributed between intervention and control groups. Data analysis will include appropriate statistical tests based on variable distribution and group comparisons.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to be conducted on patients undergoing arthroscopic surgery. The intervention group will be shown a 9,5 minute virtual reality (VR) content, created by the researcher, through VR goggles. The video content will be recorded by the researcher and a team using an Insta360 Pro device. The content will be a simulation involving healthcare professionals in various roles. The footage will be taken from the patient's perspective.

Once the operating room introduction video is completed, expert opinions will be gathered from 10 professionals in the field. Among the experts, 2 will be academicians, 2 will be experienced operating room nurses with at least 10 years of experience, 2 will be orthopedic surgeons, 1 will be a patient who has undergone arthroscopic surgery, 1 will be an anesthesiologist, and 1 will be an anesthesia technician. If the validity index from expert feedback is at least 80%, the video will be finalized.

Before the training content is shown, the VR goggles will be sanitized using an appropriate antiseptic solution, and then placed on the patient. The training content will consist of a 3D operating room introduction video. The device to be used for this training is a portable VR headset developed by Meta. It offers an advanced VR experience with its Snapdragon XR2 Gen 2 processor and high-resolution screens. Additionally, the device complies with the European Union's CE marking requirements and the Federal Communications Commission (FCC) regulations in the United States.

The introduction video will feature a patient's perspective and will detail the entire process up until the administration of anesthesia. During the video, the nurse will provide simultaneous narration, which will be heard by the patient through headphones. The content of the video will cover processes such as the patient's exit from the hospital room, transfer to the operating room, surgical safety procedures, introduction of devices used in surgery, prevention of pressure ulcers and hypothermia, and monitoring stages. The nurse will remain with the patient throughout the training.

After the training content is shown, measurements will be taken using the scales at specified time intervals. The study will compare the differences in surgical fear, anxiety levels, physiological parameters, pain levels, and satisfaction between the control group and the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years
* Patients scheduled for arthroscopic surgery
* Those who have not undergone any previous surgical procedures
* Patients who will undergo surgery under general anesthesia
* Individuals without communication barriers
* Patients with clear consciousness, and orientation to person, place, and time
* Those with no neurological or psychiatric disorders
* Individuals with no severe visual or auditory impairments

Exclusion Criteria:

* Inability to communicate with the patients
* Development of a life-threatening health problem after surgery
* Transition to open surgery during the procedure
* Patients who wish to withdraw from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety level: State-Trait Anxiety Inventory - STAI | STAI trait:1 day before surgery, prior to intervention/education STAI state:1.Immediately after STAI-II measurement 2.Immediately after the intervention/education 3.On the day of surgery, prior to premedication 4.Within 2 hours after surgery
  State-Trait Anxiety Inventory (STAI-I and STAI-II): This inventory measures individuals' current (state) anxiety levels and general (trait) anxiety tendencies. Both forms consist of 20 items and use a 4-point Likert-type response scale.
  Score range: Varies between 20 and 80. Higher scores: Indicate higher anxiety levels. Lower scores: Indicate lower anxiety levels.

SECONDARY OUTCOMES:
Surgical fear level: Measured using the Surgical Fear Scale | 1. Immediately after STAI-I measurement, 2. Immediately after the intervention/education, 3.On the day of surgery, prior to premedication
  The change in surgical fear levels in the intervention and control groups will be assessed. Surgical Fear Scale (SFS); scores range from 0 to 100, with higher scores indicating greater fear.

OTHER OUTCOMES:
Pain level: Measured using the Numeric Rating Scale (NRS) | Pain levels will be recorded within the first 2 hours after surgery using the NRS.
  This measure will compare the postoperative pain levels between the virtual reality education and standard education groups. Pain level will be assessed using the Numerical Rating Scale (NRS).
  Minimum Value: 0 (No Pain) Maximum Value: 10 (Worst Pain) Higher Scores: Indicate worse outcomes, meaning more severe pain.
Physiological parameters: Measured using electrodermal activity (EDA), heart rate, blood pressure (systolic and diastolic), respiratory rate, and peripheral oxygen saturation (SpO2). | Before the intervention, immediately after the intervention, 20 minutes before the transfer to the operating room on the morning of surgery, and 15 minutes after arriving at the inpatient ward.
  This measure will assess the physiological responses (electrodermal activity, heart rate, blood pressure, respiratory rate, and SpO2) in patients after virtual reality education and standard education
Satisfaction | Satisfaction will be measured within 2 hours after discharge procedures have started.
  Patient satisfaction will be assessed using a satisfaction scale. Satisfaction with the intervention will be assessed using the Satisfaction Scale.
  Minimum Value: 1 (Very Dissatisfied) Maximum Value: 10 (Very Satisfied) Higher Scores: Indicate better outcomes, meaning higher satisfaction levels.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem Atasehir Hospitla, Istanbul, Ataşehir
  - Acibadem Altunizade Hospital, Istanbul, ataşehir

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data through open access in the relevant journal, after anonymizing the data. No personally identifiable information will be included, and only anonymized data will be shared. We plan to make the data accessible on the journal's data platform after the publication date of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Start Date: 01.01.2026 (When the publication process begins) End Date: 01.07.2026 (6 months after publication)

REFERENCES:
- [Background] Ugras GA, Kanat C, Yaman Z, Yilmaz M, Turkmenoglu MO. The Effects of Virtual Reality on Preoperative Anxiety in Patients Undergoing Colorectal and Abdominal Wall Surgery: A Randomized Controlled Trial. J Perianesth Nurs. 2023 Apr;38(2):277-283. doi: 10.1016/j.jopan.2022.07.005. Epub 2022 Oct 29. PMID 36319521
- [Background] Gursoy A, Candas B, Guner S, Yilmaz S. Preoperative Stress: An Operating Room Nurse Intervention Assessment. J Perianesth Nurs. 2016 Dec;31(6):495-503. doi: 10.1016/j.jopan.2015.08.011. Epub 2016 May 6. PMID 27931701
- [Background] Delaney LD, Clauw DJ, Waljee JF. The Management of Acute Pain for Musculoskeletal Conditions: The Challenges of Opioids and Opportunities for the Future. J Bone Joint Surg Am. 2020 May 20;102 Suppl 1(Suppl 1):3-9. doi: 10.2106/JBJS.20.00228. No abstract available. PMID 32251126
- [Background] Morgan H, Nana M, Phillips D, Gallagher S. The Effect of a VIrtual RealiTy Immersive Experience Upon Anxiety Levels, Procedural Understanding, and Satisfaction in Patients Undergoing CArdiac CaTHeterization: The VIRTUAL CATH Trial. J Invasive Cardiol. 2021 Sep;33(9):E681-E686. doi: 10.25270/jic/20.00664. Epub 2021 Aug 8. PMID 34398809
- [Background] Rizzo MG Jr, Costello JP 2nd, Luxenburg D, Cohen JL, Alberti N, Kaplan LD. Augmented Reality for Perioperative Anxiety in Patients Undergoing Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2329310. doi: 10.1001/jamanetworkopen.2023.29310. PMID 37589975
- [Background] Cheng JYJ, Wong BWZ, Chin YH, Ong ZH, Ng CH, Tham HY, Samarasekera DD, Devi KM, Chong CS. Preoperative concerns of patients undergoing general surgery. Patient Educ Couns. 2021 Jun;104(6):1467-1473. doi: 10.1016/j.pec.2020.11.010. Epub 2020 Nov 21. PMID 33303283
- [Background] Chan SL, Sit JWH, Ang WW, Lau Y. Virtual reality-enhanced interventions on preoperative anxiety symptoms in adults undergoing elective surgery: A meta-analysis and meta-regression. Int J Nurs Stud. 2024 Dec;160:104886. doi: 10.1016/j.ijnurstu.2024.104886. Epub 2024 Aug 30. PMID 39270596
- [Background] Ugras GA, Yildirim G, Yuksel S, Ozturkcu Y, Kuzdere M, Oztekin SD. The effect of different types of music on patients' preoperative anxiety: A randomized controlled trial. Complement Ther Clin Pract. 2018 May;31:158-163. doi: 10.1016/j.ctcp.2018.02.012. Epub 2018 Feb 17. PMID 29705448
- [Background] Ruiz Hernandez C, Gomez-Urquiza JL, Pradas-Hernandez L, Vargas Roman K, Suleiman-Martos N, Albendin-Garcia L, Canadas-De la Fuente GA. Effectiveness of nursing interventions for preoperative anxiety in adults: A systematic review with meta-analysis. J Adv Nurs. 2021 Aug;77(8):3274-3285. doi: 10.1111/jan.14827. Epub 2021 Mar 23. PMID 33755246
- [Background] Leland DP, Pareek A, Therrien E, Wilbur RR, Stuart MJ, Krych AJ, Levy BA, Camp CL. Neurological Complications Following Arthroscopic and Related Sports Surgery: Prevention, Work-up, and Treatment. Sports Med Arthrosc Rev. 2022 Mar 1;30(1):e1-e8. doi: 10.1097/JSA.0000000000000322. PMID 35113840